CLINICAL TRIAL: NCT04637815
Title: A Social Network AOD Intervention for Homeless Youth Transitioning to Housing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, David Kennedy, Senior Social / Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RHINO Study ID: 2018-0539; R34DA047502 (NIH)
Record Dates: First submitted 2020-11-10; First posted 2020-11-20 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will consist of four sessions spaced two weeks apart that will last approximately 30 minutes each and consist of two parts: a network interview to capture network data about the time period since their last interview and a discussion of a resulting network visualization conducted in a motivational interviewing style. Participants will receive the intervention as part of existing case management.
  Interventions: Behavioral: Motivational Network Intervention
- Usual Care (Active Comparator): As part of residency, participants receive regular case management meetings.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Motivational Network Intervention — Every 2 weeks, residents attend meetings with their case manager. These meetings are customized to the needs of the resident at the time of the meeting. Participants randomized into the Motivational Network Intervention arm are offered an additional discussion about their social networks. Case managers ask participants to answer a series of standardized questions about people they know. After these questions are answered, case managers show participants a series of images representing these answers. While showing these images, case mangers engage the participant in discussions about what they notice using Motivational Interviewing techniques. The goal is to discuss what the participant wants to change and state strategies about achieving these changes.
  Arms: Intervention
Other: Usual Care — Residents attend regular case management meetings with their case managers as a condition of their residency in the housing program. These sessions are customized do the needs of the resident at the time of the meeting. Participants randomized into the usual care arm will be offered these sessions every 2 weeks.
  Arms: Usual Care

SUMMARY:
This project will pilot test a computer-assisted social network intervention, using motivational interviewing techniques, that can help case managers work with formerly homeless young adults who recently transitioned to supportive housing to reduce substance use and increase permanent supportive connections during this critical transitional period.

DETAILED DESCRIPTION:
The goal of this study is to conduct a pilot evaluation of a motivational network intervention (MNI) to reduce substance use and strengthen supportive connections for recently homeless 18-25 year-olds who have transitioned to a housing program. The goal of this pilot study is to evaluate, through a small randomized controlled trial (Stage 1b), the added benefit of incorporating the MNI into case management for transitional age youth (TAY) residents of housing programs. We hypothesized that residents receiving the MNI as part of case management would show more positive changes in their substance use behaviors and the composition and structure of their personal networks (i.e., greater proportion of network members who are low-risk) over a 3-month follow-up period compared to residents receiving usual case management only.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25
* In a housing program for homeless transition age youth
* Past month substance use
* Screen positive for past-year harmful substance use

Exclusion Criteria:

• Not able to speak/understand English

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Village Family Services, Burbank, California, United States

REFERENCES:
- [Derived] Kennedy DP, Osilla KC, Tucker JS. Feasibility of a computer-assisted social network motivational interviewing intervention to reduce substance use and increase supportive connections among emerging adults transitioning from homelessness to housing. Addict Sci Clin Pract. 2022 May 3;17(1):26. doi: 10.1186/s13722-022-00307-4. PMID 35505383
- [Derived] Tucker JS, Kennedy DP, Osilla KC, Golinelli D. Motivational network intervention to reduce substance use and increase supportive connections among formerly homeless emerging adults transitioning to housing: study protocol for a pilot randomized controlled trial. Addict Sci Clin Pract. 2021 Mar 16;16(1):18. doi: 10.1186/s13722-021-00227-9. PMID 33726809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through a nonprofit agency in Los Angeles County that provides a comprehensive continuum of care to transitional age youth experiencing homelessness. The agency's case managers offered eligibility screening to all residents who had been at the facility for less than one year. Residents who consented to be contacted by the study team completed an eligibility screener and provided contact information and informed consent if eligible and willing to participate.
Pre-assignment Details: Recruitment was delayed throughout the project due to COVID-19 social-distancing restrictions and frequent resident quarantines. These restrictions also limited the number of MNI sessions that could be scheduled and completed. During the final year of the project, the project team ended randomization and assigned all study participants to the CONNECT arm to adjust for recruitment/session delivery shortfalls.
Groups:
- Intervention: The intervention will consist of four sessions spaced two weeks apart that will last approximately 30 minutes each and consist of two parts: a network interview to capture network data about the time period since their last interview and a discussion of a resulting network visualization conducted in a motivational interviewing style. Participants will receive the intervention as part of existing case management.
  Motivational Network Intervention: See earlier description
- Usual Care: As part of residency, participants receive regular case management meetings. Since we are interested in evaluating the added benefit of the MNI over usual case management, residents in the control condition will be asked to meet with their case manager four times (once every two weeks) during their participation in the study. These meetings are anticipated to last approximately 30-60 minutes and will be customized to the residents' needs.
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 26 | 13
Completed | 20 | 11
Not Completed | 6 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis participants include all those who completed baseline surveys. Case managers recruited and provided informed consent to 39 eligible and interested participants. A separate interviewer subsequently contacted and completed the baseline interview with the participant by telephone. 3 eligible participants never completed the baseline interview and are not part of the analysis population because they never provided any responses to any questions necessary for measures.
Groups:
- Usual Care: As part of residency, participants receive regular case management meetings.
  Usual Care: See earlier description
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 24 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 12 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.2 (2.4) | 21.7 (1.7) | 21.3 (2.17)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 12 | 6 | 18
  Unspecified | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 4 | 17
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 2 | 3 | 5
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 11 | 2 | 13
Number of Days Cannabis Used [Mean (Standard Deviation); unit: days] | 4.79 (5.76) | 5.67 (8.67) | 5.08 (6.75)
Proportion of Risky Network Members [Mean (Standard Deviation); unit: proportion] | .24 (.27) | .05 (.07) | .164 (.222)
Number of Drinks Consumed on Drinking Days [Mean (Standard Deviation); unit: drinks per day] | 3.75 (5.45) | 3.58 (2.78) | 3.69 (4.68)
Number of Drinking Days [Mean (Standard Deviation); unit: days] | 4.79 (5.76) | 5.67 (8.67) | 5.08 (6.75)
Number of Days Consumed 5 (for Men) or 4 (for Women) Drinks on a Single Occasion [Mean (Standard Deviation); unit: days] | 2.63 (5.24) | 4.17 (8.33) | 3.14 (6.36)
Proportion of Supportive Network Members [Mean (Standard Deviation); unit: proportion] | .56 (.31) | .60 (.30) | .59 (.30)
Average network centrality - risky alters [Mean (Standard Deviation); unit: average connections] — Participants listed names of network contacts ("alters"). Risky alters are defined as those they used more alcohol or drugs with than usual. Participants also listed how many other alters each alter knew. The measure "connections" was calculated for each alter to indicate the number of other network members they knew.
  For each respondent, average connections was calculated for different types of network members, including "risky alters". The average connection measure was calculated by adding up "connections" for each "risky alter" and dividing it by the overall number of alters.
  average connections | .328 (.401) | .167 (.30) | .271 (.372)
Average network centrality - supportive alters [Mean (Standard Deviation); unit: average connections] — Participants listed names of network contacts ("alters"). Supportive alters are defined as those who provide at least one type of support. Participants also listed how many other alters each alter knew. The measure "connections" was calculated for each alter to indicate the number of other network members they knew.
  For each respondent, average connections was calculated for different types of network members, including "supportive alters". The average connection measure was calculated by adding up "connections" for each "supportive alter" and dividing it by the overall number of alters.
  average connections | 1.50 (1.31) | 2.24 (2.65) | 1.77 (1.89)

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Cannabis Used
Description: Count of days that respondent used cannabis in the past 30 days
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 11
days | 23.7 (10.5) | 7.36 (11.2)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Equivalence — t-tests for continuous variables and chi-squared tests for categorical variables; t-test, 2 sided — Statistical threshold of significance is .05; We also conducted difference in differences (DID) analysis by first constructing measures of difference between follow-up and baseline for each participant for each measure and then comparing the means of these difference measures for each arm

2. Primary Outcome: Proportion of Risky Network Members
Description: Proportion of network members who engaged in substance use or the participant used more substances when they were with the network member.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: proportion of network members
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 11
proportion of network members | .242 (.342) | .0797 (.106)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Equivalence — t-tests for continuous variables and chi-squared tests for categorical variables; t-test, 2 sided — Statistical threshold of significance is .05; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Number of Drinks Consumed on Drinking Days
Description: Participants reported on the typical number of drinks they consumed on drinking days in the past month.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: drinks per day
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 11
drinks per day | 2.30 (2.25) | 3.64 (5.54)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Equivalence — t-tests for continuous variables and chi-squared tests for categorical variables; t-test, 2 sided — Statistical threshold of significance is .05; [other analysis details as in outcome 1, analysis 1]

4. Primary Outcome: Number of Drinking Days
Description: Number of days in the past month (0-30) that participants reported engaging in any alcohol use.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 11
days | 7.45 (8.47) | 6.09 (9.35)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Equivalence — t-tests for continuous variables and chi-squared tests for categorical variables; t-test, 2 sided — Statistical threshold of significance is .05; [other analysis details as in outcome 1, analysis 1]

5. Primary Outcome: Number of Days Consumed 5 (for Men) or 4 (for Women) Drinks on a Single Occasion
Description: Number of days in the past month (0-30) that participants reported engaging in heavy alcohol use (5 or more drinks for men and four or more drinks for women on a single occasion).
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 11
days | 1.95 (2.89) | 2.91 (8.35)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Equivalence — t-tests for continuous variables and chi-squared tests for categorical variables; t-test, 2 sided — Statistical threshold of significance is .05; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 3 months, from the time they are screened / recruited by case managers until they complete the follow-up assessment. Each participant is offered 4 sessions separated by 2 weeks each. After they complete the final session with their case manager, they are contacted about completing their final assessment. During this time, project staff discuss any adverse events for participants who have been screened until they complete follow-up interviews with case managers during weekly project meetings.
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/12
Other Adverse Events (participants affected / at risk) | 0/24 | 0/12

LIMITATIONS AND CAVEATS:
Recruitment was delayed throughout the project due to COVID-19 social-distancing restrictions and frequent resident quarantines. These restrictions also limited the number of MNI sessions that could be scheduled and completed. During the final year of the project, the project team ended randomization and assigned all study participants to the CONNECT arm to adjust for recruitment/session delivery shortfalls. The resulting study sample was underpowered to detect intervention effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT04637815/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT04637815/ICF_001.pdf